CLINICAL TRIAL: NCT02517385
Title: Multicenter Prospective Uncontrolled Non-comparative Open Interventional Clinical Study of Phase III for Assessment of the Safety and Effectiveness of Using the Drug Phosphatidylcholine Paste 600 mg in Patients With Acute and Chronic Liver Diseases and Clinical Symptoms of Dysfunction of the Gastrointestinal Tract During 12-week Therapy Course
Brief Title: Essentiale® Paste in Patients With Gastrointestinal Symptoms in Acute or Chronic Liver Diseases
Acronym: EPLID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHOLIL06301; U1111-1131-0460 (Other: UTN)
Record Dates: First submitted 2015-07-20; First posted 2015-08-07 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Hepatic and Hepatobiliary Disorders
MeSH Terms: conditions — Digestive System Diseases | interventions — Phosphatidylcholines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phosphatidylcholine paste (Experimental): One dose of phosphatidylcholine paste 600 mg given orally 3 times a day at Days 0, 28, 56, and 84
  Interventions: Drug: Phosphatidylcholine

INTERVENTIONS:
Drug: Phosphatidylcholine — Pharmaceutical form:Paste Route of administration: Oral

SUMMARY:
Primary Objective:

To assess safety of Phosphatidylcholine paste 600 mg (ESSENTIALE® paste) oral 3 times a day for 12 weeks in patients with gastrointestinal symptoms in acute and chronic liver diseases.

Secondary Objectives:

To assess effectiveness on symptomatic improvement in patients with gastrointestinal symptoms in acute and chronic liver diseases.

To monitor compliance.

DETAILED DESCRIPTION:
The total study duration per patient will be 13 weeks that consists of 1-week pre-screening period and a 12-week treatment period.

ELIGIBILITY:
Inclusion criteria:

* Males and females ≥18 years of age and less than 66 years old.
* Patients with gastrointestinal symptoms (fatigue, abdominal pain/discomfort, early satiety, fullness discomfort after meal, nausea/vomiting, belching/abdominal distension, at least one rated as "Moderate Problem" or higher severity at screening visit) in acute and chronic liver diseases receiving conventional treatment for the underlying pathology.
* Before entering the study, patients will be advised to stop alcohol intake and must agree not to consume alcohol and undergo alcohol withdrawal program, diet control, and exercise program.
* The patient is able and willing to undertake all study required procedures and has the ability to take oral medications.
* Patients with nonalcoholic fatty liver disease (NAFLD) diagnosed by ultrasound examination in absence of severe fibrosis as per Investigator's judgment.
* Diagnosis of acute or chronic viral hepatitis as manifested by a combination of the following symptoms: jaundice (acute viral hepatitis), dark-colored urine (acute viral hepatitis), light-colored stools (acute viral hepatitis), pruritus, pruritic red hives, fever, nausea, vomiting, anorexia, aversion to smoking and right upper abdominal discomfort, pain or feeling of pressure, with abnormal alanine aminotransferase (ALT) (approximately 1.5 x upper limit of normal [ULN]).
* Patient has given written informed consent.
* Fertile patients must agree to use an acceptable method of contraception to avoid pregnancy for the duration of the study:
* Total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to study drug administration).
* Vasectomized partner of female subjects.
* Hormonal contraceptives.
* Double-barrier method (condoms and diaphragm or vaginal cap plus spermicidal sponge, jellies, or cream).
* Intrauterine Device (IUD).

Exclusion criteria:

* Patients <18 years of age and >66 years old.
* Female patient of childbearing potential without negative pregnancy test.
* Breastfeeding woman.
* Hypersensitivity to phosphatidylcholine or any substance of the product.
* Patient is known to be human immunodeficiency virus (HIV) positive.
* Congenital lack of α-1 antitrypsin.
* Gastroesophageal Reflux Disease (GERD).
* Autoimmune hepatitis.
* Fulminant hepatitis.
* Severe steatohepatitis: transaminases level is beyond 5 times upper normal range.
* Previous liver biopsy that demonstrated greater than or equal to 15% steatosis.
* Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dL, total bilirubin >1.5 mg/dL, or prothrombin time/international normalized ratio >1.3 times normal at screening, or history or presence of ascites or encephalopathy, or bleeding from esophageal varices.
* Diagnosis of cancer.
* Parenteral nutrition.
* Advanced liver disease (eg, ascites, bleeding esophageal varices, hepatic encephalopathy, cancer or hepatic metastasis).
* History of other serious chronic liver disease, including serious metabolic diseases, documented by appropriate test(s).
* Evidence of upper abdomen organic serious diseases (ulcer, etc.).
* Platelet count <130 000 cells/mm^3.
* Serum creatinine level >1.5 times the upper limit of normal at screening, or creatinine clearance <60 cc/min, or currently on dialysis.
* History of drug abuse within a year prior to Day 0.
* Current or recent use (within 15 days of screening) of any hepatoprotector drug.
* Use of warfarin, metronidazole, or chronic use of acetaminophen/paracetamol greater than three grams per day.
* Use of oral steroids within 30 days prior to screening.
* Use of concomitant medication disturbing the liver function or CYP3A4 inducers.
* Patients who have taken drugs able to induce fatty liver for over 3 months within 1 year of participation in this study; (ie, amiodarone, tamoxifen, methotrexate, tetracyclines, glucocorticoids, over usual dose of estrogen for hormone replacement therapy, valproate, St. John's Wort, etc.).
* Patients who have taken any medications that could affect the treatment for nonalcoholic steatohepatitis: insulin, insulin sensitizer (ie, metformin, thiazolidinedione, high dose of vitamin E, high dose of ursodeoxycholic acid, pentoxifylline, S-adenosyl methionine, betaine, types of statin, types of fibrate, orlistat, etc.).
* History of solid organ or bone marrow transplantation.
* History and current immunologically mediated disease (eg, inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hepatitis, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis, polyorganic pathology) that could affect inflammatory biomarkers.
* History and current thyroid disease poorly controlled on prescribed medications.
* History and current significant renal, endocrine, cardiac, or pulmonary disease.
* Other serious liver diseases or systemic pathologies (malignancies, central nervous system). Some examples are severe hypertension, morbid obesity (body mass index >40), severe mental illness, diabetes type 1, and poorly controlled diabetes type 2.
* Other conditions which, in the Investigator's opinion, make the patient unsuitable for enrollment (such as coronary artery disease or active gastrointestinal conditions that might interfere with drug absorption).
* The patient is currently participating in any clinical trial (marketed product or otherwise) or has done so within 30 days prior to screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Frequency (number) of adverse events (AEs) related to the investigational drug | Week 12

SECONDARY OUTCOMES:
Change from baseline in patient percentage of global overall symptoms using Likert Scale | Weeks 4, 8, and 12
Change from baseline in gastrointestinal symptom percentage score | Weeks 4, 8, and 12
Percentage of patients with AEs regardless of the Investigator's assessment of relationship to the investigational drug | Weeks 4, 8, and 12
Number of AEs regardless of the Investigator's assessment of relationship to the investigational drug | Weeks 4, 8, and 12
Number of patients who complied with the prescribed treatment | Weeks 4, 8, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Moscow, Russia